CLINICAL TRIAL: NCT03033628
Title: Pain Perception of Maxillary Infiltration Injection of Dental Local Anesthesia Using "DentalVibe Comfort System" Compared to Maxillary Infiltration Injection Alone in a Group of Egyptian Children: A Randomized Clinical Trial
Brief Title: Pain Perception of Dental Local Anesthesia Using "DentalVibe Comfort System" in a Group of Egyptian Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Muaaz Marwan halal, principal investigator, Cairo University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CEBC-CU-2017-01-06
Record Dates: First submitted 2017-01-22; First posted 2017-01-27 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Dental Anxiety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- DV group (Experimental): Device: injection using DentalVibe comfort system. giving maxillary infiltration dental local anesthesia with the aid of "DentalVibe comfort system" on one side of the maxillary arch prior extraction of primary molar tooth
  Interventions: Device: injection using DentalVibe comfort system
- C group (Active Comparator): Device: traditional dental injection giving maxillary infiltration dental local anesthesia without the aid of "DentalVibe comfort system" on the other side of the maxillary arch prior extraction of primary molar tooth
  Interventions: Device: traditional dental injection

INTERVENTIONS:
Device: injection using DentalVibe comfort system — giving maxillary infiltration injection of dental local anesthesia using DentalVibe comfort system.
  Arms: DV group
Device: traditional dental injection — giving maxillary infiltration injection of dental local anesthesia without using DentalVibe comfort system.
  Arms: C group

SUMMARY:
The aim of this study is to compare pain during maxillary infiltration local anesthesia injection with the aid of DentalVibe comfort system in comparison to maxillary infiltration injection alone in pediatric dental patients.

DETAILED DESCRIPTION:
The aim of this study is to compare pain during maxillary infiltration local anesthesia injection with the aid of DentalVibe comfort system in comparison to maxillary infiltration injection alone.

Intervention:

History taking from the child and the parent including personal, medical and dental history as in the examination sheet (Appendix A) to assess inclusion criteria.

Clinical procedure:

Intervention group:

Clinical examination using mirror and probe to assess inclusion criteria. Before initiating the treatment, the site of the injection will be dried then prepped with antiseptic solution swab, then a topical anaesthetic agent (topical anesthetics 20% benzocaine) will be applied with a cotton tip applicator for 60 sec.

Demonstration will be performed by putting the device into direct contact with the children's nails before applying the device intraorally.

The cheek will be retracted and the device will be turned on.

1mL of local anesthetic solution (articaine hypochloride 4% with 1:100.000 epinephrine, Septodont) will be injected using a 27 gauge needle which will be delivered over 1 min.

Control group:

AS that of the intervention group except, the device will be used only as a cheek retractor during the injection, but will be turned off.

Assessment:

Objective assessment will be performed by observing the patients behavior using the FLAAC scale during the anesthetic injection and needle insertion.

Subjective evaluation will be obtained using the Wong-Baker FACES pain rating scale.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy children aged 6-7 years old.
2. Apparently healthy Children.
3. Cooperative children.
4. Children with carious maxillary bilateral primary molars indicated for extraction.

Exclusion Criteria:

1. Children who are allergic to amide group.
2. Children with Neurologic disorders.
3. Children with mental disability.
4. Presence of periapical or gingival legion.
5. Severe Gingivitis.

Ages: 6 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 21 (Estimated)
Dates: Start 2017-04-01 (Estimated); Primary Completion 2017-06-01 (Estimated); Study Completion 2018-01-01 (Estimated)

PRIMARY OUTCOMES:
pain during injection | within 1 year
  pain assessment using FLACC behavioral pain assessment (scale 0-10) and Wong-Baker FACES pain rating scale (scale 0-10) e 0: Relaxed and comfortable 1-3: Mild discomfort. 4-6: Moderate pain. 7-10: Severe discomfort or pain or both.

CONTACTS AND LOCATIONS:
Overall Officials: Norhan El-dokky, PHD, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No